CLINICAL TRIAL: NCT03053479
Title: Comparison of the Efficacy of Three Surgical Methods in the Treatment of POP: Sacrocolpopexy,the Amreich-Richter Procedure and Transvaginal Mesh
Brief Title: Comparison of the Efficacy of Sacrocolpopexy, the Amreich-Richter Procedure and Transvaginal Mesh
Acronym: SAME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamil Svabik, MD PhD, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAME
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: surgery; native tissue prolapse repair; laparoscopic sacrocolpopexy; vaginal mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic sacrocolpopexy (Experimental): Laparoscopic sacrocolpopexy will be performed in the following way: Identification of the promontory, dissection of the peritoneum above the promontory and preparation of the ligamentum longitudinale anterior, peritoneum dissection, dissection of the vesicovaginal septum up to the bladder neck, dissection of the rectovaginal septum towards the perineum, application of Y mesh, fixation to the vaginal apex using non-absorbable sutures, and for anterior and posterior vaginal wall absorbable sutures. Fixation of the upper mesh arm to the ligamentum longitudinale anterior using non-absorbable suture, following with complete peritoneum closure above the mesh. The procedure could include salpingo-oophorectomy, supracervical hysterectomy or total hysterectomy (concomitant procedures are not exclusion criteria).
  Interventions: Procedure: Laparoscopic sacrocolpopexy
- Transvaginal mesh procedure (Experimental): Hydrodissection of the anterior vaginal wall, midline anterior colporrhaphy, preparation beyond the endopelvic fascia, mesh kit with bilateral fixation to sacrospinous ligaments should be used. The procedure could include salpingo-oophorectomy, total hysterectomy and posterior vaginal wall repair (concomitant procedures are not exclusion criteria).
  Interventions: Procedure: Transvaginal mesh procedure
- Amreich-Richter procedure: (Experimental): At least unilateral fixation with non-absorbable suture to sacrospinous ligament (fixation could be performed from the anterior approach). At the time of anterior vaginal wall repair or traditional posterior approach, it is possible to use a device for stich fixation (for example Capio, I- stitch etc). The procedure could include salpingo-oophorectomy, total hysterectomy and posterior vaginal wall repair (concomitant procedures are not exclusion criteria).
  Interventions: Procedure: Amreich-Richter procedure

INTERVENTIONS:
Procedure: Laparoscopic sacrocolpopexy — see arm/group descriptions
  Arms: Laparoscopic sacrocolpopexy
Procedure: Transvaginal mesh procedure — see arm/group descriptions
  Arms: Transvaginal mesh procedure
Procedure: Amreich-Richter procedure — see arm/group descriptions
  Arms: Amreich-Richter procedure:

SUMMARY:
Pelvic organ prolapse, POP, is a common health problem affecting up to 40% of women. Very little is known about the factors associated with surgical failure. Studies have identified a variety of risk factors: younger age, high body mass index and advanced preoperative prolapse (grade III-IV) have been associated with an increased risk of reoperation in some studies. According to some studies patients had poorer anatomical outcome after traditional repairs but were able to enjoy the same quality of life as after transvaginal mesh surgery or laparoscopic sacrocolpopexy. The purpose of this study is to assess and compare the efficacy of these three procedures in a randomized controlled trial.

DETAILED DESCRIPTION:
Pelvic organ prolapse, POP, is a common health problem affecting up to 40% of women. The lifetime likelihood of undergoing at least one incident of pelvic organ prolapse surgery has been estimated at approximately 13%. The prevalence of reoperation after primary pelvic reconstructive surgery is high at around 30%, while some studies report the figure as up to 58%. In the early 1990s the perception of pelvic floor defects and urinary incontinence in women started to change significantly. The diagnostics and management of these defects became an independent uro-gynecological sub-specialization within gynaecology and obstetrics, and it has been included among 4 basic sub-specializations recognized by the European Board and College of Obstetrics and Gynecology. Surgical treatment is indicated in women with symptomatic POP when conservative management has failed or has been declined. There is no indication for repair of asymptomatic POP as an isolated procedure where surgical correction is of uncertain benefit and adds peri- and post-operative risks. The objective of our treatment should always aim to restore quality of life and comfort. Very little is known about the factors associated with surgical failure. Studies have identified a variety of risk factors: younger age, high body mass index and advanced preoperative prolapse (grade III-IV) have been associated with an increased risk of reoperation in some studies, while other studies did not prove these hypotheses. One factor which significantly influences the result of the pelvic organ surgery is the presence of pelvic floor injury. Injury of the musculus levator ani mainly affects the results of traditional vaginal wall repair, with 60% risk of recurrence. In the last few years, in an attempt to reduce recurrence and improve the outcome of reconstructive surgery in the treatment of pelvic organ prolapse, surgeons have started to use transvaginally introduced prosthetic material (mesh). This type of surgery significantly increases the efficacy of the procedure (anatomic cure rate over 90%), but its use is associated with a risk of some complications (vaginal erosions and potential consecutive infections, granulomas, dyspareunia, vesico-vaginal fistulas, chronic pain) thereby potentially reducing patient quality of life and leading to additional surgery. If the mesh is introduced during sacrocolpopexy and the vaginal wall is not open, there is a significant decrease of mesh-related complications. Laparoscopic sacrocolpopexy is considered the gold standard for the management of apical prolapse with high long-term efficacy. According to some studies patients had poorer anatomical outcome after traditional repairs but were able to enjoy the same quality of life as after transvaginal mesh surgery or laparoscopic sacrocolpopexy. Therefore the investigators plan to assess the efficacy in a randomized trial of three different surgical methods (the Amreich-Richter procedure, transvaginal mesh and laparoscopic sacrocolpopexy) in patients with high risk of recurrence; i.e. patients with advanced pelvic organ prolapse (at least stage III) and proved injury of pelvic floor muscles.

Aims of the study: To evaluate on the basis of a prospective randomized trial the clinical efficacy of three different surgical procedures (the Amreich-Richter procedure, transvaginal mesh and laparoscopic sacrocolpopexy) in women with advanced pelvic organ prolapse and proved pelvic floor muscle injury

All patients will undergo complete urogynecological investigation before the procedure (history, clinical examination, assessment of pelvic organ prolapse using the POPQ system, examination of the levator resting tone and contraction (Oxford scale),where appropriate urodynamics according to ICS recommendation and ultrasound examination), and they will fill in standardized international questionnaires (ICIQ-UI SF, PISQ 12, UDI_POPDI-CRADI, POP-SF). Ultrasound examinations will be performed as a combined examination using a convex probe, from abdominal and perineal approaches, and sectoral vaginal probe from the introital approach. Investigation will be preserved mainly in digital form and partly on videotapes. Acquired data from 4D imagery will be preserved in the form of data set and processed with appropriate software. Ultrasound examination will assess standards parameters describing position of the urethrovesical junction, bladder descent, uterus descent, posterior vaginal wall descent (rectocele, enterocele). Using 3D/4D ultrasound examination the status of the pelvic floor will be evaluated (presence of avulsion of puborectalis muscle, abnormal genital hiatus distension). Women will be randomized into three groups: 1. Group - Laparoscopic sacrocolpopexy 2. Group - Transvaginal mesh procedure 3. Group - Amreich-Richter procedure (traditional vaginal wall repair with apical fixation to sacrospinous ligament.

All surgical procedures will be performed under general, spinal or epidural anesthesia where indicated, and antibiotic prophylaxis will be used. Surgery will be provided in standardized steps, see arm descriptions.

In an early postoperative check-up 2-3 weeks after surgery evaluation of post-operative pain will be performed and late post-operative complication such as de novo constipation, urinary retention, infections analyzed. The next post-operative complete examination is planned for 3 months after surgery (the same examination as before the procedure including clinical exam, ultrasound the QoL (ICIQ- SF, POP-SF, PISQ 12, UDI_POPDI-CRADI, TS-VAS). The next visits will be provided one year and two years after surgery, and the procedure will be the same as at the 3-month check-up. In addition to pre-operative ultrasound examination the position of the mesh will be monitored. All patients in this study will have a minimum one year follow-up and, whenever possible, a two year follow-up. Postoperative follow-up will be terminated if the result of surgery is evaluated as a failure, and in these cases reoperation will be offered. Further post-operative follow-up up to five years is also planned.

ELIGIBILITY:
Inclusion Criteria:

* age over18
* signed informed consent
* symptomatic pelvic organ prolapse stage III or higher (according to the International Continence Society Pelvic Organ Prolapse quantification system - POPQ) in anterior and apical (central) compartments, one at least stage II and the second at least stage III
* presence of at least a unilateral avulsion injury of the puborectalis muscle
* agreement with postoperative follow-up.

Exclusion Criteria:

* previous pelvic reconstructive surgery with mesh
* isolated posterior compartment prolapse
* previous radiotherapy in true pelvis
* contraindication for one of the planned surgical methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | 2 years
  absence of pelvic organ prolapse (using the POPQ system - maximal I. stage prolapse)
Number of failures in each group | 2 years
  failure is defined as pelvic organ prolapse stage II or higher using the POPQ system during the clinical examination, or as a descent 1 cm below the lower edge of pubic bone based on ultrasound examination.
de novo dyspareunia | 2 years
  new occurence of painful sexual intercourse after the surgery.
mesh related complications | 2 years
  extrusion rate, pain

SECONDARY OUTCOMES:
Change of the genital hiatus size | 2 years
  Measured at Valsalva from rendered 4D volume
Distance of mesh from the bladder neck | 2 years
  Measured from sagittal plane, transperineal ultrasound
Lowest position of the mesh | 2 years
  Measured from sagittal plane, transperineal ultrasound at Valsalva. Distance in relation to a horizontal line at the level of symphysis.
ICIQ-UI SF | 2 years
  International Consultation on Incontinence questionnaire, urinary incontinence, short form
POP-SS | 2 years
  Pelvic organ prolapse symptom scale
PISQ-12 | 2 years
  Prolapse/incontinence sexual questionnaire
PFDI | 2 years
  Pelvic floor distress inventory
TS-VAS | 2 years
  Treatment satisfaction - visual analog scale
de novo stress urinary incontinence | 2 years
  any occurence
de novo symptoms of overactive bladder | 2 years
  any occurence
reoperation for pelvic organ prolapse recurrence | 2 years
  rate

CONTACTS AND LOCATIONS:
Locations (7):
- Czechia (6):
  - Frýdek-Místek regional hospital, Frýdek-Místek
  - Faculty of Medicine in Olomouc, Palackeho University, Olomouc
  - Faculty of Medicine in Pilsen, Charles University, Pilsen
  - General University Hospital, 1st Faculty of Medicine, Charles University, Prague
  - Hospital Na Bulovce, 1st Faculty of Medicine, Charles University, Prague
  - Tomas Bata Regional Hospital in Zlin, Zlín
- Louis Pasteur University Hospital Kosice, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No
IPD sharing not planned